CLINICAL TRIAL: NCT00890227
Title: Incidence of Proximal Junctional Kyphosis (PJK) in Long Posterior Spinal Fusion: A Prospective Controlled Randomized Study Comparing Traditional Open Surgery to Minimally Invasive Percutaneous Technique at the Proximal Fusion Levels/Levels
Brief Title: Incidence of Proximal Junctional Kyphosis (PJK) in Long Posterior Spinal Fusion: A Study Comparing Traditional Open Surgery to Minimally Invasive Percutaneous Technique at the Proximal Fusion Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NA_00002729; SORC_KMK_08_006 (Other: JHU SOM Spine Outcomes Research Center)
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Scoliosis; Kyphosis
Keywords: scoliosis; kyphosis; Surgical treatment
MeSH Terms: conditions — Scoliosis; Kyphosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional technique (Active Comparator): All level open instrumented posterior spinal fusions
  Interventions: Procedure: Traditional technique
- Minimally invasive technique (Active Comparator): Open surgery for all the levels except the proximal segment (most proximal instrumented level) where minimally invasive technique will be used.
  Interventions: Procedure: Minimally invasive technique

INTERVENTIONS:
Procedure: Traditional technique — All level open instrumented posterior spinal fusions
  Arms: Traditional technique
Procedure: Minimally invasive technique — Open surgery for all the levels except the proximal segment (most proximal instrumented level) where minimally invasive technique will be used.
  Arms: Minimally invasive technique

SUMMARY:
This research is being done to compare two methods of surgery to treat scoliosis and/or kyphosis of the spine.

DETAILED DESCRIPTION:
Currently, there are two different surgical methods used in the treatment of these problems. One method includes an all open posterior spinal fusion (large incision with opening of the muscles); this is also known as a traditional technique. The second method involves an open surgery for the portion of the spine requiring a fusion except the very top area, where minimally invasive technique (smaller incision and without opening of the muscles) is used.

One possible side effect of either method for surgical repair is a condition called proximal junctional kyphosis (PJK). PJK occurs in the form of fracture at the top vertebra involved in the surgery or as a loss of correction of spinal alignment achieved, through gradual bending forward of the spine over time. In this study we want to compare the rate of PJK between two groups of patients undergoing long posterior spinal instrumentation fusion.

People undergoing long posterior spinal instrumented fusion may join.

About 68 people will join.

ELIGIBILITY:
Inclusion Criteria:

* Individuals presenting for surgical correction of scoliosis and/or kyphosis of the thoracolumbar spine are the primary target for enrollment.
* Men and women ages 18 years or older will be eligible for participation in the current study.
* In addition, individuals must be able to provide informed consent (Mini-Mental State Examination score of at least 18/30).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
To estimate the rate of proximal junctional fracture or instrumentation failure leading to kyphosis and loss of correction between two groups. | 12 months
  rate of proximal junctional fracture or instrumentation failure

SECONDARY OUTCOMES:
To evaluate complication rate between the two groups. | 3 months
  rate of complications
To compare the total operative time between the two groups of surgical patients (as stratified above). | 12 months
  operative time
To compare the length of hospital stay between the two groups of surgical patients (as stratified above). | 12 months
  length of hospital stay
To compare the total recovery time between the two groups of surgical patients (as stratified above). | 12 months
  total recovery time
To assess change in self-reported pain following surgery between two groups of surgical patients (as stratified above). | 12 months
  pain rating
To assess change in self-reported functional limitations following surgery between two groups of surgical patients (as stratified above). | 12 months
  oswestry disability index

CONTACTS AND LOCATIONS:
Overall Officials: Khaled M Kebaish, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Outpatient Center, Baltimore, Maryland, United States